CLINICAL TRIAL: NCT06333457
Title: Presence and Relapse Rates in Patients With Alcohol Use Disorder Using Virtual Reality
Acronym: PRE-VR
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alva Lütt, Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA4/024/24
Record Dates: First submitted 2024-03-17; First posted 2024-03-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VR group: 50 patients with diagnosed alcohol dependence (in-patients, patients in the outpatient department or day clinics) receiving VR Cue-Exposure Therapy (VR-CET) additional to the standard treatment.
  Interventions: Device: VR Cue-Exposure Therapy
- control group: 50 patients with diagnosed alcohol dependence (in-patients, patients in the outpatient department or day clinics) receiving standard treatment.

INTERVENTIONS:
Device: VR Cue-Exposure Therapy — Standard VR Cue Exposure Therapy (VR-CET) for the treatment of alcohol dependence
  Groups: VR group

SUMMARY:
Investigation of the influence of the sense of presence during a Virtual Reality Cue-Exposure Therapy (VR-CET) with alcohol-associated cues on craving and relapse rates.

Study group: abstinent patients (at least 18 years old) with a diagnosed alcohol dependence after completed inpatient withdrawal treatment in the the last 3 months.

Primary hypothesis: the experience of presence during a virtual presentation of alcohol in alcohol-dependent patients is associated with levels of craving for alcohol during VR-CET.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65 years
* diagnosis of alcohol dependence according to ICD-10 (F10.2)
* completed in-patient withdrawal treatment during the last 3 months
* history of alcohol craving, confrmed via craving questionnaires
* able to provide written informed consent

Exclusion Criteria:

* substance dependence other than alcohol and nicotine
* current alcohol intoxication (randomly tested via measurement of breath alcohol concentration)
* unable to understand the study information, consent form or principles of the study
* abstinence for less than 7 days or on-going consumption of alcohol
* severe neuropsychiatric disorder, e.g., schizophrenia spectrum disorders, bipolar afective disorder or substantial cognitive impairment
* somatic diseases for which VR is associated with risks, e.g. photosensitive epilepsy
* acute suicidality or acute endangerment of others
* concurrent pharmacological treatment targeting AUD (i.e. benzodiazepines) or craving (i.e. acamprosate, disulfram, naltrexone, nalmefene)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcohol dependence treated in the inpatient or outpatient psychiatric clinics or day clinics of the Psychiatric University Hospital Charité at St. Hedwig-Hospital/ Department of Psychiatry and Neurosciences Campus Charité Mitte/ Theodor-Wenzel Werk Berlin / Jüdisches Krankenhaus Berlin / Vivantes Auguste-Viktoria-Klinikum
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Craving | VR-group: 6 appointments/6 weeks. Every appointment pre, during (approx. 20 min VR exposure) and post VR exposure / control group: 6 appointments/6 weeks, measures once every appointment, both groups: follow up appointments after 6 weeks + after 12 weeks
  subjective craving for alcohol, measured with Visual Analogue Scales (VAS; 0 - 10 with higher scores indication higher craving levels)
Craving | VR-group: 6 appointments/6 weeks. Every appointment pre and post VR exposure / control group: 6 appointments/6 weeks, measures once every appointment, both groups: follow up appointments after 6 weeks + after 12 weeks
  subjective craving for alcohol, measured with Alcohol Urge Questionnaire (AUQ; scores ranging from 8-56, higher scores indicating higher craving levels)
Craving | VR-group: 6 appointments/6 weeks. Every appointment pre VR exposure / control group: 6 appointments/6 weeks, measures once every appointment, both groups: follow up appointments after 6 weeks + after 12 weeks
  subjective craving for alcohol, measured with Obsessive Compulsive Drinking Scale (OCDS, scores 0-56; higher scores indicating higher craving levels)

SECONDARY OUTCOMES:
Relapse rates | both groups: follow up appointment after 6 weeks, follow up appointment after 12 weeks
  TLFB (timeline followback method) for assessment of individual's alcohol intake
Quality of Life | both groups: assessment during appointment 1 and 6 and during follow up appointments after 6 and 12 weeks
  Assessment of quality of life via WHOQOL-BREF questionnaire, 0-100% (higher scores indicating better quality of life)
Motion Sickness | VR group: pre and post VR exposure (6 appointments/6 weeks)
  Assessment of VR motion sickness using the Simulator Sickness Questionnaire (SSQ; scores from 0-48, higher scores indicating more side effects)
Presence in VR | VR group: post VR exposure (6 appointments/6 weeks)
  Igroup Presence Questionnaire (IPQ; score range from 0 to 84, with higher scores indicating more realistic perceptions)

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Charité at St. Hedwig Hospital, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided